CLINICAL TRIAL: NCT00561756
Title: Phase I Trial to Assess Safety and Immunogenicity of Xenogeneic CD20 DNA Vaccination With Patients With B-Cell Lymphoma
Brief Title: Vaccine Therapy in Treating Patients With Recurrent B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-100; MSKCC-07100
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma
Keywords: cutaneous B-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; recurrent marginal zone lymphoma; recurrent mantle cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Flow Cytometry; Immunoenzyme Techniques

ARMS (1):
- Vaccine Therapy (Experimental): This single arm, open-label, phase I clinical trial of xenogeneic CD20 DNA vaccination is designed to evaluate its safety in patients with B cell lymphoma. The study is a dose escalation study at three test doses, 0.5 mg, 2 mg and 4 mg of purified plasmid DNA per injection. There will be an initial cohort of three patients receiving a pre-level 1 dose of 0.1 mg/vaccination before proceeding to the three test doses.
  Interventions: Biological: plasmid DNA vaccine therapy; Other: flow cytometry; Other: immunoenzyme technique

INTERVENTIONS:
Biological: plasmid DNA vaccine therapy
Other: flow cytometry
Other: immunoenzyme technique

SUMMARY:
RATIONALE: Vaccines made from mouse DNA may help the body build an effective immune response to kill cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of mouse DNA vaccine in treating patients with recurrent B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and feasibility of intramuscular DNA vaccination with a plasmid DNA vector expressing the mouse extracellular domain of CD20, namely pINGmminiCD20. Doses of pING-mminiCD20 will be escalated by group to determine the optimal biological dose.

Secondary

* To evaluate antibody and T-cell responses to CD20 after vaccination.
* To observe patients for evidence of any antitumor response generated after vaccination.

OUTLINE: The entire immunization schedule comprises five injections administered every three weeks (for a total of approximately four and one half months). After the second injection, blood will be drawn for assessment of antibody and T-cell responses. After the fifth and final injection, blood will again be drawn for assessment of antibody and T-cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a functional immune system as determined by the following tests:
* Serum proteins immunoelectrophoresis (serum IgG levels ≥ 0.5 g/dL are required)
* No evidence of anergy as shown by positive skin test with tetanus toxoid, mumps or Candida. OR
* Circulating T-cells as measured by flow cytometry (serum CD4+ and CD8+ T-cell counts ≥ 250 and 150 cells/μL, respectively) Patients must have histologically proven (and confirmed at MSKCC) B-cell lymphoma of any histology, excluding Burkitt's lymphoma, Lymphoblastic lymphoma (due to their aggressiveness and low likelihood of response to immune therapy).
* CD20 surface expression must be confirmed by immunohistochemical staining or flow.
* Measurable disease is not a pre-requisite for enrollment in the study. However, if a patient does have measurable disease as evidenced by imaging studies, these have to be done within eight weeks of starting treatment.
* Patients must have a Karnofsky performance status ≥ 70%.
* Patients with evidence of active disease, progression of disease or relapsed disease following one or more prior regimens of chemotherapy, immunotherapy or radiation therapy (including autologous stem cell transplants), not requiring immediate cytoreductive chemotherapy. All treatment must be completed at least four weeks prior to administration of the first vaccination, except immunotherapy and radioimmunotherapy, which must be completed at least 90 days prior to receiving the first vaccination. Active disease includes patients with minor or partial responses after therapy as evidenced by FDG-avid disease or biopsy.
* Age ≥ 18.
* Adequate contraception during study enrollment.
* Avoidance of breast-feeding their infants during the study enrollment.
* Patients must have adequate organ and marrow function as defined below:
* Absolute Neutrophil Count ≥ 1,000/uL
* Platelets ≥ 75,000/uL
* Total bilirubin ≤ 2.5 times institutional upper limit
* AST/ALT ≤ 2.5 times institutional upper limit
* Creatinine ≤ 2 mg/dL
* PT/PTT ≤ 1.5 times institutional upper limit
* Patients must have no signs of congestive heart failure according to the New York Heart Failure Guidelines Class III/IV.

Exclusion Criteria:

* Patients who have had chemotherapy or radiation therapy within 4 weeks prior to entering the study.
* Patients who have undergone an allogeneic stem cell transplant at any time.
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who have received immunotherapy (i.e. rituximab) or radioimmuno therapy (i.e. tositumomab or ibritumomab) within the past 90 days.

Patients who display signs of anergy as indicated by skin testing.

* Patients with Burkitt's lymphoma and Lymphoblastic Lymphoma.
* Patients who have been previously immunized with any type of DNA vaccine.
* Patients who have positive anti-DS-DNA antibodies.
* Patients with life expectancy less than 3 months from the time of enrollment.
* Patients with serious underlying medical conditions, active infections requiring the use of antimicrobial drugs or active bleeding.
* Patients with active Hepatitis C (HC) or Hepatitis B (HB) infection, the latter defined as a positive test for HBsAg or measurable viral load. In patients who are HBsAg negative but HBsAg positive (regardless of HBsAb status), a HB viral load will be performed and if positive the subject will be excluded. If the subject is HBsAg negative, HBcAb positive (regardless of HBsAb status) but with negative HBV viral load, the subject may be included but must undergo HBV DNA PCR testing at least every two months from the start of treatment during the routine study visits for as long as the subject remains on study. Prophylactic antiviral therapy, in addition to the monitoring described above, may be initiated at the discretion of the investigator.

Patients with documented HIV infection or other immunodeficiency disorder or on chronic steroids treatment.

* Patients with autoimmune diseases such as but not limited to rheumatoid arthritis, Sjogren disease, ulcerative colitis, autoimmune hepatitis.
* Pregnant or nursing women. Women of child-bearing age will be tested for qualitative β-HCG within 2 weeks of immunization.
* Patients receiving other investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity | 2 years

SECONDARY OUTCOMES:
Antibody and T-cell responses against CD20 | 2 years
Antitumor response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: M. Lia Palomba, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Andrew D. Zelenetz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Alan N. Houghton, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States